CLINICAL TRIAL: NCT05851274
Title: Transradial Access for Ruptured Intracranial Aneurysms Embolization--A Multicentre, Randomised, Open-label,Non-inferiority Trial
Brief Title: Transradial Access for Ruptured Intracranial Aneurysms Embolization
Acronym: TRA-RIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Lu Hua, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRA-RIA
Record Dates: First submitted 2023-04-12; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Transradial Access
Keywords: transradial access; ruptured intracranial aneurysms; intervention

STUDY DESIGN:
Intervention Model Description: In the experimental group, the transradial access (TRA) was used, which was to puncture the radial artery and insert a radial sheath to establish a surgical pathway for embolization of the aneurysm; In the control group, transfemoral access (TFA) was used to embolize the aneurysms, which was to puncture the femoral artery and insert the femoral sheath to establish a surgical pathway for embolizing the aneurysm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transradial access (Experimental): In this group, the transradial access (TRA) was used, which was to puncture the radial artery and insert a radial sheath to establish a surgical pathway for embolization of the aneurysm.
  Interventions: Procedure: transradial access
- Transfemoral access (Active Comparator): In this group, transfemoral access (TFA) was used to embolize the aneurysms, which was to puncture the femoral artery and insert the femoral sheath to establish a surgical pathway for embolizing the aneurysm.
  Interventions: Procedure: Transfemoral access

INTERVENTIONS:
Procedure: transradial access — In this group, the transradial access (TRA) was used, which was to puncture the radial artery and insert a radial sheath to establish a surgical pathway for embolization of the aneurysm
  Arms: Transradial access
Procedure: Transfemoral access — In this group, transfemoral access (TFA) was used to embolize the aneurysms, which was to puncture the femoral artery and insert the femoral sheath to establish a surgical pathway for embolizing the aneurysm.
  Arms: Transfemoral access

SUMMARY:
The goal of this clinical trail is to compare the difference between transradial access (TRA) and transfemoral access(TFA) for ruptured intracranial aneurysms embolization. The main question it aims to answer is: whether is TRA not inferior to TFA？ In the experimental group, the transradial access (TRA) was used, which was to puncture the radial artery and insert a radial sheath to establish a surgical pathway for embolization of the aneurysm; In the control group, transfemoral access (TFA) was used to embolize the aneurysms, which was to puncture the femoral artery and insert the femoral sheath to establish a surgical pathway for embolizing the aneurysms.The two groups of patients received an oral loading dose of aspirin (300mg) plus clopidogrel (300mg) on the day of surgery, while patients who were unable to take orally were given nasal feeding. During the operation, systemic heparinization was performed with a starting dose of 75U/kg intravenous injection, and the injection was halved every 1h until 1000U. After the operation, protamine neutralizing heparin (1mg protamine neutralizing 100U heparin) was used.

ELIGIBILITY:
Inclusion Criteria:

1. The age is between 18 and 75 years old.
2. Receiving interventional embolization treatment for intracranial aneurysms.
3. CT scan of the skull shows subarachnoid hemorrhage, and CTA or DSA of the skull shows the presence of an intracranial aneurysm, and it is determined to be aneurysm-related subarachnoid hemorrhage after evaluation by a neurosurgical specialist.
4. At least one side of the bilateral radial arteries can be used to establish surgical access.
5. Evaluation of radial artery patency: Barbeau test type A-C .
6. Hunt-Hess grade 1-3, Glasgow coma score ≥ 8.
7. Agreed to participate in this study and willing to cooperate with follow-up. -

Exclusion Criteria:

1. Preoperative upper limb ultrasound or DSA showed radial artery spasm and arteriovenous fistula.
2. Artery CTA or DSA showed vascular anatomical abnormalities such as axillary artery occlusion, and acute angle between the left common carotid artery and the subclavian artery, which may affect the operation.
3. The patient's condition is serious and may die or remain in a coma after surgery, as assessed by a specialist.
4. Received radial or femoral artery puncture examination or treatment within 1 month.
5. The patient refused to participate in the study or cooperate with follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2023-05-10 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
The success rate of operation | during the procedure
  The success rate of operation

SECONDARY OUTCOMES:
Incidence of ischemic events | immediately after the procedure
  Incidence of ischemic events
Incidence of hemorrhage events | immediately after the procedure
  Incidence of hemorrhage events

CONTACTS AND LOCATIONS:
Overall Officials: Hua L Lu Hua, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chivot C, Bouzerar R, Yzet T. Transitioning to Transradial Access for Cerebral Aneurysm Embolization. AJNR Am J Neuroradiol. 2019 Nov;40(11):1947-1953. doi: 10.3174/ajnr.A6234. Epub 2019 Oct 3. PMID 31582386
- [Result] Chen SH, Snelling BM, Shah SS, Sur S, Brunet MC, Starke RM, Yavagal DR, Osbun JW, Peterson EC. Transradial approach for flow diversion treatment of cerebral aneurysms: a multicenter study. J Neurointerv Surg. 2019 Aug;11(8):796-800. doi: 10.1136/neurintsurg-2018-014620. Epub 2019 Jan 22. PMID 30670622
- [Result] Chiu AH. Is Transradial Access a Replacement Technique for Transfemoral Access in Neurointervention? AJNR Am J Neuroradiol. 2021 Mar;42(3):493-494. doi: 10.3174/ajnr.A6935. Epub 2021 Jan 14. No abstract available. PMID 33446496